CLINICAL TRIAL: NCT00725946
Title: A Pilot Study to Determine Radioiodide Accumulation and Dosimetry in Breast Cancers Using 124I PET/CT
Brief Title: Pilot Study to Determine Radioiodide Accumulation and Dosimetry in Breast Cancers Using 124I PET/CT
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Irene L. Wapnir, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRS0001; 98583 (Other: Stanford University Alternate IRB Approval Number); SU-03142008-1044 (Other: Stanford University); IRB-11927 (Other: Stanford Universtiy)
Record Dates: First submitted 2008-07-09; First posted 2008-07-31 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer; Breast Cancer Early Stage Breast Cancer (Stage 1-3); Breast Cancer Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Iodine-124

ARMS (1):
- Iodine-124 PET-CT scan (Experimental)
  Interventions: Drug: Iodine-124; Radiation: PET/CT with Iodine-124

INTERVENTIONS:
Drug: Iodine-124
Radiation: PET/CT with Iodine-124

SUMMARY:
This is a pilot imaging study for women whose tumors express NIS [Na+I- symporter, sodium iodide symporter]. Eligibility is limited to the presence of strong (3+) and/or plasma membrane staining in > 20% of cells as determined by immunohistochemical methods. A total of 10 patients will be imaged with 124I PET/CT (serial scans over 24 hour period) to determine radioiodide uptake and distribution in tumor tissue. Thyroid iodide uptake and retention will be blocked beginning one week prior to 124I PET/CT scan with thyroid hormone (T3) and methimazole (impedes organification). Tumor, organ and whole body dosimetry will be calculated in each patient.

ELIGIBILITY:
Inclusion Criteria:1. Stage I-IV breast cancer. Patients must have clinical or radiographic evidence of localized or metastatic disease.

2. Criteria for NIS-positivity are defined as: >= 20% of cells with plasma membrane and/or strong intracellular/plasma membrane immunoreactivity 3. Any previous therapy including radiation therapy is allowable. 4. Women 18 years of age or older. 5. Patients must have a life expectancy of at least 3 months 6. Patients with ECOG Performance Status 0-3 will be eligible. 7. If on chemotherapy, thyroid suppression should be initiated no sooner than two weeks after last chemotherapy cycle.

8. Ability to understand and willingness to sign a written informed consent document.

9. Discontinuation of hormonal or biological therapies for the 10 days of the study is preferred but not mandated.

10. Laboratory tests (CBC, comprehensive metabolic panel) must be performed within 120 day prior to study initiation. Exclusion Criteria:1. History of metastatic thyroid cancer 2. Exclude the use of cytotoxic, hormonal or biological agents for one week prior to and during imaging.

3. Pregnant or nursing patients will be excluded from the study as iodide can accumulate in the breast and is transported across the placenta.

4. Inability to tolerate thyroid hormone and/or methimazole pre-imaging treatment.

5. History of thyroid cancer (because patient could have concomitant thyroid cancer metastases and therefore competitively concentrate radioiodides) 6. Psychiatric or addictive disorders that are not adequately controlled and would preclude obtaining informed consent.

7. Patients with heart disease or other significant cardiac risk factors will be excluded from receiving thyroid suppressive therapy so as to avoid precipitating a cardiac arrhythmia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Radioiodide accumulation | 2 years
  To evaluate radioiodide accumulation in women with immunohistochemically NIS (Na+/I- symporter)-positive breast cancers using 124I PET/CT.

SECONDARY OUTCOMES:
Dosimetry | 2 years
  To calculate dosimetry in tumor, thyroid and whole body.

CONTACTS AND LOCATIONS:
Overall Officials: Irene L. Wapnir, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States